CLINICAL TRIAL: NCT03604666
Title: Ambulatory Process of Elderly Patient for Skin and Breast Cancer Surgery
Brief Title: Follow-up of Elderly Patients in Ambulatory Surgery
Acronym: PAPA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: K170702J
Record Dates: First submitted 2018-06-10; First posted 2018-07-27 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2018-05

CONDITIONS: Breast Cancer; Skin Cancer; Surgery; Ambulatory
Keywords: Breast Cancer; Skin cancer; Surgery; Ambulatory
MeSH Terms: conditions — Breast Neoplasms; Skin Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Health care process with Nurse Navigator: A Nurse Navigator will:
  * Be present at the announcement consultation
  * Give information on the outpatient circuit
  * Offer assistance for patients over 75 years
  * Complete onco-geriatric orientation questionnaires
  * Take care of patients on the ambulatory circuit
  Interventions: Other: Health care process with Nurse Navigator
- Health care process: Health care process

INTERVENTIONS:
Other: Health care process with Nurse Navigator — A Nurse Navigator will:
  * Be present at the announcement consultation
  * Give information on the outpatient circuit
  * Offer assistance for patients over 75 years
  * Complete onco-geriatric orientation questionnaires
  * Take care of patients on the ambulatory circuit
  Groups: Health care process with Nurse Navigator

SUMMARY:
The number of surgical procedures performed in ambulatory hospitalization for cancers of the skin or breast is increasing for medical and economic reasons. But the protocols of care and the clinical pathways are poorly adapted for elderly patients with physical or cognitive impairment.

The goal of this study is to test the impact of an oncology ambulatory surgical care in patients aged 75 years or older, with breast or skin cancer and treated in Henri Mondor hospital on the increase in the proportion of patients operated on an outpatient basis

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 75 years old with breast cancer or skin cancer and requiring surgical excision: partial mastectomy, lumpectomy, axillary dissection, cutaneous excision, etc.
* With an indication of ambulatory care
* Patient (legal representative or trusted person or member of the family) having been informed and having given his non-oral objection to his participation in the study
* Possessing a health insurance

Exclusion Criteria:

* Patients reserved for breast reconstruction to the operative gesture of tumor resection.
* Patients do not consent to care because of deficient mental state.
* Formal surgical contraindication due to a pathology medical device does not allow anesthesia. - Participation in another interventional research or be in the exclusion period after a previous search, if applicable

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over 75 years consulting at the dermatological crossroads or "crossroads breast" and requiring surgery for a cancer of the skin or breast (without reconstruction)
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients operated on an outpatient basis | 3 month
  Test the impact of an oncology ambulatory surgical care in patients aged 75 years or older, with breast or skin cancer and treated in Henri Mondor hospital

SECONDARY OUTCOMES:
Number of death | at Day 30 and Day 90
  Test the impact of the new organization of care on the mortality
Number of patients converted to conventional care | at Day 30 and Day 90
  Test the impact of the new organization of care on the proportion of patients converted to conventional care
Number of the passage to emergencies | at Day 30 and Day 90
  Test the impact of the new organization of care on the passage to emergencies
Number of not programmed hospitalizations | at Day 30 and Day 90
  Test the impact of the new organization of care on the not programmed hospitalizations
The autonomy Activities of Daily Living (ADL) | at Day 30 and Day 90
  Test the impact of the new organization of care on the autonomy (ADL/IADL)
The autonomy Instrumental Activities of Daily Living (IADL) | at Day 30 and Day 90
  Test the impact of the new organization of care on the autonomy (ADL/IADL)
Number of institutionalization to Long-term care and skilled nursing facilities | at Day 30 and Day 90
  Test the impact of the new organization of care on the institutionalization to Long-term care and skilled nursing facilities
Number of passage to Long-term care and skilled nursing facilities | at Day 30 and Day 90
  Test the impact of the new organization of care on the passage to Long-term care and skilled nursing facilities
Number of postoperative complications | at Day 90
  Test the impact of the new organization of care on the postoperative complications
Costs of care | at Day 30 and Day 90
  Test the impact of the new organization of care on the costs of care
Patients' satisfaction (questionnaire) for the prospective part of the study | at Day 30 and Day 90
  Test the impact of the new organization of care on patients' satisfaction
Patient's quality of life (EQ50 questionnaire, for the prospective part of the study) | at Day 30 and Day 90
  Test the impact of the new organization of care on quality of life (EQ50) (for the prospective part of the study)

CONTACTS AND LOCATIONS:
Overall Officials: Romain BOSC, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Bosc, Créteil, France

IPD SHARING:
Plan to Share IPD: No